CLINICAL TRIAL: NCT00540839
Title: A Phase III Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Prospectively Evaluate Efficacy of Montelukast in Patients Aged 6 Months to 5 Years With Chronic Asthma
Brief Title: A Study of Montelukast (MK-0476) Compared With Fluticasone in Pediatric Participants With Chronic Asthma (MK-0476-303)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on input from regulatory agencies, it is not necessary to conduct this study. An ongoing study was sufficient for regulatory purposes.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0476-303; 2007_583 (Other: Telerx ID Number)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma | interventions — montelukast; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Experimental): Participants receive montelukast 4 mg oral granules (OG) or 4 mg chewable tablets (CT) once daily (QD) for 24 weeks and placebo to fluticasone 50 mcg inhalation aerosol twice daily (BID) for 24 weeks. Participants aged >6 months to <2 years receive montelukast 4 mg packet of OG QD for 24 weeks. Participants aged >2 years to <64 months receive montelukast 4 mg CT QD for 24 weeks.
  Interventions: Drug: Montelukast sodium; Drug: Placebo to fluticasone
- Fluticasone (Active Comparator): Participants receive fluticasone 50 mcg inhalation aerosol twice daily (BID) for 24 weeks and placebo to montelukast 4 mg QD for 24 weeks. Participants aged >6 months to <2 years receive placebo packet of OG QD for 24 weeks. Participants aged >2 years to <64 months receive placebo CT QD for 24 weeks.
  Interventions: Drug: Placebo to montelukast; Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Montelukast sodium — Montelukast 4 mg OG or montelukast 4 mg CT
  Other Names: MK-0476; Singulair®
  Arms: Montelukast
Drug: Placebo to montelukast — Placebo OG or CT
  Arms: Fluticasone
Drug: Fluticasone propionate — Fluticasone 50 mcg inhalation aerosol metered dose inhaler
  Arms: Fluticasone
Drug: Placebo to fluticasone — Placebo inhalation aerosol metered dose inhaler
  Arms: Montelukast

SUMMARY:
A study to determine the effects of montelukast (MK-0476) on pediatric participants with chronic asthma compared with fluticasone. The primary hypotheses are that, over 24 weeks of treatment, montelukast will provide at least the same level of asthma control as inhaled fluticasone as measured by the percentage of days without asthma and that, over 24 weeks of treatment, daily administration of montelukast will be safe and well tolerated in children aged 6 months to 5 years with chronic asthma.

This trial was stopped at a time before any participants had actually entered the trial. Based on input from regulatory agencies, it is not necessary to conduct this study; a separate ongoing study was sufficient for regulatory purposes.

DETAILED DESCRIPTION:
This study consists of a 4-week placebo run-in period followed by a 24-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 months and 5 years, 4 months of age
* Diagnosed with asthma by a doctor
* At least 3 episodes of asthma symptoms within the last 6 months

Exclusion Criteria:

* Active or chronic breathing disease, other than asthma
* Required insertion of a breathing tube for asthma
* Major surgery within the last 4 weeks
* Currently in the hospital
* Allergic to certain drugs, and for children under 2 years of age, apples, applesauce and formula

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of days without asthma | 24 weeks
  A day without asthma is defined as a day with all of the following: no daytime symptoms, no nighttime cough, no β-agonist use, and no asthma attack (defined as a visit to a doctor, urgent care clinic, emergency room, or hospital for asthma [other than a scheduled visit to a doctor], or treatment with systemic corticosteroid during the previous 24 hours).
Number of participants who experience at least one adverse event (AE) | Up to 26 weeks
Number of participants who discontinue study drug due to an AE | Up to 24 weeks

SECONDARY OUTCOMES:
Percentage of days without daytime symptoms | 24 weeks
Percentage of days without nighttime cough | 24 weeks
Percentage of days without β-agonist use | 24 weeks

OTHER OUTCOMES:
Percentage of participants without asthma attacks | 24 weeks
Percentage of participants without corticosteroid rescues | 24 weeks
Caregiver global evaluation | Week 24
Physician global evaluation | Week 24
Percentage of days without individual daytime asthma symptoms (cough, wheeze, trouble breathing, and activity limitation) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC